CLINICAL TRIAL: NCT04053634
Title: A Multicenter, Randomized, Double-blind, Chronic-dosing, Parallel-group, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Benralizumab 100 mg in Patients With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD) With a History of Frequent COPD Exacerbations and Elevated Peripheral Blood Eosinophils (RESOLUTE)
Brief Title: Efficacy and Safety of Benralizumab in Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD) With a History of Frequent Exacerbations
Acronym: RESOLUTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3251C00014; 2019-001800-39 (EudraCT Number)
Record Dates: First submitted 2019-07-16; First posted 2019-08-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; benralizumab; Fasenra; ICS; inhaled corticosteroids; exacerbations; Lung Disease; LABA/LAMA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Administrated subcutaneously (SC) every 4 weeks for the first 3 doses, then every 8 weeks
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Administrated subcutaneously every 4 weeks for the first 3 doses, then every 8 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab solution for injection in accessorized prefilled syringe (APFS) will be administered subcutaneously (SC) every 4 weeks for the first 3 doses - Weeks 0, 4 and 8, and then every 8 weeks until the end of treatment.
  Arms: Benralizumab
Biological: Placebo — Matching placebo will be administered subcutaneously with accessorized prefilled syringe (APFS) every 4 weeks for the first 3 doses - Weeks 0, 4 and 8, and then every 8 weeks until the end of treatment.
  Arms: Placebo

SUMMARY:
Phase 3 study to evaluate the efficacy and safety of a benralizumab in patients with moderate to very severe COPD with a history of frequent COPD exacerbations and elevated peripheral blood eosinophils (≥300/μL).

Eligible patients must have a history of ≥2 moderate and/or severe COPD exacerbations in the previous year despite receiving triple (ICS/LABA/LAMA) background therapy for at least 3 months and ICS-based dual inhaled treatment for the remainder of the year. Eligible patients must also have an elevated blood eosinophil count.

The treatment period will be of variable duration and will continue until the last patient has the opportunity to complete a minimum of 56 weeks, at which point all patients will complete the study. The primary endpoint will be analyzed at Week 56.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Age 40 to 85 years
3. Male and/or female.
4. Current or former smoker with a tobacco history of ≥10 pack-years.
5. History of moderate to very severe COPD with a post-bronchodilator FEV1/FVC<0.70 and FEV1 ≤65% of predicted normal value.
6. Documented history of 2 or more COPD exacerbations that required treatment with systemic corticosteroids and/or hospitalization within 52 weeks prior to enrollment.

   1. Exacerbations treated with antibiotics alone are excluded unless accompanied by treatment with systemic corticosteroids and/or hospitalization.
   2. Hospitalization is defined as an inpatient admission ≥24 hours
   3. Previous exacerbations should be confirmed to have occurred while on stable triple therapy for COPD.
   4. At least one qualifying COPD exacerbation should occur while on stable uninterrupted triple therapy prior to enrolment.
7. Documented use of triple (ICS/LABA/LAMA) background therapy for COPD for ≥3 months immediately prior to enrollment.

   1. Treatment with at least double inhaled therapy containing ICS (e.g. ICS/LABA or ICS/LAMA) for the remaining of 52 weeks prior to enrolment. Use of LABA/LAMA is allowed if ICS cannot be tolerated.
   2. ICS in a dose approved for COPD or equivalent to ≥250 mcg of fluticasone propionate daily.
   3. Total cumulative duration of not being on double or triple background therapy must not exceed 2 months.
   4. Stable therapy/doses for the last 3 months prior to randomization.
8. Blood eosinophil count ≥300/μL at screening and documented historical eosinophil count of ≥150/μL within 52 weeks of enrollment (or repeated testing during run-in).
9. CAT total score ≥15 at Visit 1.
10. Negative pregnancy test for females of childbearing potential (WOCBP) at Visit 1.
11. Women of childbearing potential (WOCBP) must agree to use a highly effective method of birth control from enrollment throughout the study and within 12 weeks after last dose of IP.

Women not of childbearing potential are defined as women who are either permanently sterilized or postmenopausal (confirmed by FSH test for women <50 years).

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD
2. Current diagnosis of asthma, prior history of asthma or asthma-COPD overlap according to GINA/GOLD. Childhood history of asthma is allowed and defined as asthma diagnosed and resolved before the age of 18.
3. Radiological findings of a respiratory disease other than COPD contributing to respiratory symptoms. Solitary pulmonary nodules without appropriate follow up or findings of acute infection.
4. Another pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
5. Any unstable disorder that could affect patient safety, study findings or the patient's ability to complete the study.
6. Any clinically significant abnormal findings in physical examination, vital signs, ECG, laboratory tests could affect patient safety, study findings or the patient's ability to complete the study.
7. Cor pulmonale and/or right ventricular failure.
8. Long-term treatment with oxygen >4.0 L/min and/or oxyhemoglobin saturation <89% while breathing supplemental oxygen.
9. Use of any non-invasive positive pressure ventilation device (NIPPV). Note: use of CPAP for Sleep Apnea Syndrome is allowed.
10. Known immunodeficiency disorder, including positive HIV-1/2 testing.
11. Active liver disease. Chronic stable hepatitis B and C (including positive HBsAg or hepatitis C antibody testing), or other stable chronic liver disease are acceptable.
12. ALT or AST ≥3 times the upper limit of normal, confirmed by repeated testing during the run-in period.
13. Helminth parasitic infection within 24 weeks prior to enrollment, not treated or failed to respond to standard of care therapy.
14. Alcohol or drug abuse within the past year, which may compromise the study data.
15. Malignancy, current or within the past 5 years, except for adequately treated non invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma-in-situ treated with apparent success more than 1 year prior to Visit 1. Suspected malignancy or undefined neoplasms.
16. Evidence of active tuberculosis, as judged by investigator. Patients with a recent (within 2 years) first-time or newly positive PPD or Quantiferon test need to complete an appropriate course of treatment before enrollment. Evaluation will be according to the local standard of care.
17. Participation, or planned participation, in intensive COPD rehabilitation program (maintenance phase of a rehabilitation is allowed).
18. History of surgical or endoscopic lung volume reduction within the 6 months prior to enrollment. History of partial or total lung resection (single lobe or segmentectomy is acceptable).
19. Scheduled major surgical procedure during the study. Minor elective procedures are allowed.
20. History of anaphylaxis to any biologic therapy or vaccine.
21. Receipt of blood products or immunoglobulins within 30 days prior to randomization.
22. Receipt of marketed or investigational biologic product within 4 months or 5 half-lives prior to randomization, whichever is longer. Exception: Patients on stable therapy for 3 months before randomization who intend to stay on treatment throughout the study with marketed biologic products that are not likely to interfere with the safety assessment and/or efficacy of benralizumab, for example, for the treatment of osteoporosis, migraine, pain, diabetes, obesity, ocular, cardiovascular, or metabolic diseases, can participate in the study.
23. Receipt of live attenuated vaccines 30 days prior to randomization.
24. Chronic use of immunosuppressive medication or expected need for chronic use during the study.
25. Chronic use of antibiotics if duration of treatment is <9 months prior to randomization. Chronic macrolide or other antibiotic therapy is allowed provided the patient has been on stable dose/regimen for ≥9 months prior to randomization and has had ≥2 COPD exacerbations while on stable therapy.
26. Receipt of any investigational non-biologic product within 30 days or 5 half-lives prior to enrollment.
27. Receipt of benralizumab within 12 months prior to enrollment.
28. Known history of allergy or reaction to any component of the IP formulation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Annualized rate of moderate or severe COPD exacerbations | Over first 56 weeks
  Moderate or severe COPD exacerbation is defined by symptomatic worsening of COPD requiring:
  * Use of systemic corticosteroids for at least 3 days; and/or
  * Use of antibiotics; and/or
  * An inpatient hospitalization or death due to COPD

SECONDARY OUTCOMES:
Annualized rate of severe COPD exacerbations | Minimum of 1 year and an average of 2 years
  A severe COPD exacerbation is defined by symptomatic worsening of COPD requiring an inpatient hospitalization or results in death due to COPD
Annualized rate of COPD exacerbations that are associated with an emergency room/emergency department visit or a hospitalization | Minimum of 1 year and an average of 2 years
Time to first COPD exacerbation | During first 56 weeks
Change from baseline in SGRQ total and domain scores | up to 56 weeks
  St. George's Respiratory Questionnaire (SGRQ)
Change from baseline in E-RS:COPD total and domain scores | up to 56 weeks
  Evaluating Respiratory Symptoms in COPD (E-RS:COPD)
Change from baseline in pre-dose/pre-bronchodilator FEV1 | up to 56 weeks
  FEV1 is the Forced expiratory volume in one second at study site
All cause and respiratory-related mortality rate | Minimum of 1 year and an average of 2 years
Annual rate of hospitalizations due to COPD | Minimum of 1 year and an average of 2 years
Serum benralizumab concentration as a measure of pharmacokinetics | up to 56 weeks
Anti-drug antibodies (ADA) as a measure of immunogenicity | up to 56 weeks
Change from baseline in CAT total score | up to 56 weeks
  Chronic Obstructive Pulmonary Disease assessment tool (CAT)
Length of hospital stay | Minimum of 1 year and an average of 2 years
ICU (Intensive Care Unit) days | Minimum of 1 year and an average of 2 years
Annual rate of hospitalizations and emergency department visits combined | Minimum of 1 year and an average of 2 years
Annual rate of unscheduled outpatient visits including unscheduled visits to study sites | Minimum of 1 year and an average of 2 years
Annual rate of unscheduled healthcare encounters | Minimum of 1 year and and average of 2 years

OTHER OUTCOMES:
Safety and tolerability of benralizumab in patients with moderate to very severe COPD | Minimum of 1 year and average of 2 years
  AEs, vital signs, clinical laboratory, and ECG

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University School of Medicine, 3401 North Broad Street, Suite 745 PP, Philadelphia, PA 19140
Locations (304):
- United States (80):
  - Research Site, Surprise, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Palm Springs, California
  - Research Site, Westminster, California
  - Research Site, Stamford, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pensacola, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Michigan City, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Georgetown, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Toms River, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New Windsor, New York
  - Research Site, The Bronx, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Elizabeth City, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, DuBois, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Abingdon, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Williamsburg, Virginia
  - Research Site, Everett, Washington
  - Research Site, Spokane, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Cudahy, Wisconsin
- Argentina (11):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autónoma de Buenos Aire
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Australia (5):
  - Research Site, Caringbah
  - Research Site, Melbourne
  - Research Site, South Brisbane
  - Research Site, Southport
  - Research Site, Spearwood
- Austria (6):
  - Research Site, Bad Ischl
  - Research Site, Bludenz
  - Research Site, Feldbach
  - Research Site, Grieskirchen
  - Research Site, Linz
  - Research Site, Thalheim
- Belgium (2):
  - Research Site, Edegem
  - Research Site, Erpent
- Brazil (9):
  - Research Site, Blumenau
  - Research Site, Botucatu
  - Research Site, Florianópolis
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Bulgaria (3):
  - Research Site, Kozloduy
  - Research Site, Rousse
  - Research Site, Stara Zagora
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, St. John's, NF
  - Research Site, Ajax, Ontario
  - Research Site, Barrie, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Stouffville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Chicoutimi
- Chile (5):
  - Research Site, Chile
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
- China (24):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Ganzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hebei
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
- Colombia (6):
  - Research Site, Barranquilla
  - Research Site, Cali
  - Research Site, Floridablanca
  - Research Site, Medellín
  - Research Site, Pereira
  - Research Site, Zipaquirá
- Czechia (5):
  - Research Site, Brandýs nad Labem
  - Research Site, Jindřichův Hradec
  - Research Site, Ostrava
  - Research Site, Rokycany
  - Research Site, Teplice
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Odense C
  - Research Site, Roskilde
  - Research Site, Vejle
- Germany (14):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Koblenz
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, Neu-Isenburg
  - Research Site, Peine
  - Research Site, Potsdam
  - Research Site, Rheine
  - Research Site, Warendorf
- Greece (4):
  - Research Site, Athens
  - Research Site, Exohi Thessaloniki
  - Research Site, Ioannina
  - Research Site, Thessaloniki
- Hungary (12):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Encs
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Komárom
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Törökbálint
- India (7):
  - Research Site, Calicut
  - Research Site, Coimbatore
  - Research Site, Guntur
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Thane
  - Research Site, Vijayawada
- Italy (7):
  - Research Site, Cona
  - Research Site, Genoa
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (27):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Himeji-shi
  - Research Site, Hitachi-Naka
  - Research Site, Joyo-shi
  - Research Site, Kawachinagano-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kure-shi
  - Research Site, Matsusaka-shi
  - Research Site, Mizunami-shi
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sagamihara-shi
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Seto-shi
  - Research Site, Shinagawa-ku
  - Research Site, Toshima-ku
  - Research Site, Toyonaka-shi
  - Research Site, Ueda-shi
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, Veracruz
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Leeuwarden
- New Zealand (4):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Dunedin
  - Research Site, Hamilton
- Philippines (4):
  - Research Site, Iloilo City
  - Research Site, Los Baños
  - Research Site, Marilao
  - Research Site, Quezon City
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Chęciny
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wieluń
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Laredo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santander
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Göteborg
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Stockholm
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Mersin
- United Kingdom (13):
  - Research Site, Barnsley
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Bradford
  - Research Site, Chertsey
  - Research Site, Cottingham
  - Research Site, Leicester
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Perth
  - Research Site, Southampton
  - Research Site, Stockton-on-Tees
  - Research Site, Wishaw
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hồ Chí Minh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: This is a poster on the Resolute study. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3251C00014&attachmentIdentifier=e179b7eb-c2d8-4b45-ad4d-14aef6dbee7a&fileName=RESOLUTE_Poster.pdf&versionIdentifier=